CLINICAL TRIAL: NCT04110275
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of Thrombolytic Therapy With Recombinant Human Tissue-type Plasminogen Activator Derivative for Acute Pulmonary Embolism
Brief Title: Injection of Recombinant Human Tissue-type Plasminogen Activator Derivative for Acute Pulmonary Embolism(rPA)
Acronym: rPA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angde Biotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD-RTL-203
Record Dates: First submitted 2019-09-24; First posted 2019-10-01 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Acute Pulmonary Embolism
Keywords: Acute Pulmonary Embolism
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Masking Description: observers are masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose group (Experimental): Recombinant human tissue-type plasminogen activator derivative(rPA) for injection: 18 mg, Intravenous injection for 2 minutes or more.
  A separate venous access should be used for bolus injection,a common venous access shared with other drugs is not allowed for injection. And no other drugs mixed with test drug during the injection.
  Interventions: Drug: Recombinant human tissue-type plasminogen activator derivative
- high dose group (Experimental): Recombinant human tissue-type plasminogen activator derivative (rPA) for injection: the first injection of 18 mg rPA is pushed slowly for 2 minutes or more,the second injection of 9mg rtPA is pushed for 1 minute or more.The interval between the two injections should be controlled accurately about 30 minutes.
  A separate venous access should be used for bolus injection,a common venous access shared with other drugs is not allowed for injection. And no other drugs mixed with test drug during the injection.
  Interventions: Drug: Recombinant human tissue-type plasminogen activator derivative
- comparative group (Active Comparator): Recombinant tissue plasminogen activator for injection: continuous intravenous injection for 2 hours.
  Interventions: Drug: Recombinant human tissue-type plasminogen activator

INTERVENTIONS:
Drug: Recombinant human tissue-type plasminogen activator derivative — Recombinant human tissue-type plasminogen activator derivative(rPA,chemical name: Reteplase,brand name:Ruitongli) 18mg/10ml/stick, provided by AngDe Biotech Pharmaceutical Co.,LIMITED(LTD)
  Other Names: Ruitongli
  Arms: high dose group; low dose group
Drug: Recombinant human tissue-type plasminogen activator — Recombinant human tissue-type plasminogen activator(rt-PA,chemical name:Alteplase,brand name: Actilyse)50mg/stick,provided by Boehringer Ingelheim Pharma Gesellschaft mit beschrankter Haftung(GmbH)&Co,
  Other Names: Actilyse
  Arms: comparative group

SUMMARY:
The purpose of this trial is to compare the efficacy and safety of Recombinant Human Tissue-Type Plasminogen Activator Derivative(rPA) and Recombinant Tissue-Type Plasminogen Activator(rt-PA) for the treatment of acute pulmonary embolism.

This trial includes two stages, the first stage is to study the dosage of administration of the test drug(rPA), the second is to compare the efficacy and safety of rPA and rt-PA. Both of the two stages are randomized, open and parallel controlled.

DETAILED DESCRIPTION:
This trial is a multicenter, randomized, open and parallel controlled project designed for patients with acute pulmonary embolism requiring thrombolysis after anticoagulant therapy in high-risk and middle-high risk populations.

For the first stage: Subjects who are qualified for the screening criteria according to the inclusion and exclusion criteria will be randomly assigned to low-dose test drugs, high-dose test drugs or reference drugs for thrombolytic therapy at a ratio of 1:1:1.

For the second stage: Subjects who are qualified for the screening criteria according to the inclusion and exclusion criteria will be randomly assigned to rPA(test group)or rt-PA(control group) for thrombolytic therapy at a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk acute pulmonary embolism: the main manifestations are shock and hypotension.Systemic systolic blood pressure <90 millimetre of mercury (mmHg) (1mmHg=0.133kPa), or a decrease from the base value ≥40 millimetre of mercury for more than 15min.
* Patients with moderate to high-risk acute pulmonary embolism who have worsened anticoagulant therapy require thrombolytic therapy:

(Patients with moderate to high-risk acute pulmonary embolism: Right ventricular dysfunction (RVD) and elevated cardiac biomarkers coexist.)

1. RVD diagnostic criteria: imaging evidence including echocardiography or CT:1) Ultrasound examination is consistent with the following performance: 1. right ventricular dilatation (right ventricular end-diastolic diameter / left ventricular end-diastolic diameter > 1.0 or 0.9); 2. right ventricular free wall movement amplitude decreased; 3. tricuspid regurgitation speed increased; 4. tricuspid annulus systolic displacement decreased (<17mm); 2) Computed Tomographic Pulmonary Angiography examination meets the following conditions: right ventricular dilatation (right ventricular end-diastolic diameter / left ventricular end-diastolic diameter > 1.0 or 0.9) found at the four-chamber heart level;
2. Cardiac biological markers including N terminal pro B type natriuretic peptide (NT-proBNP/BNP) and troponin elevation;

Diagnostic criteria for worsening after anticoagulant therapy in patients with moderate to high risk acute pulmonary embolism:

Hemodynamic deterioration (defined as meeting at least one of the following conditions: 1. requires cardiopulmonary resuscitation; 2. systemic systolic blood pressure <90 mmHg (1 mmHg = 0.133 kPa), or a decrease in basal value ≥ 40 mmHg for more than 15 min, or with terminal Low organ perfusion (limb cold or urine volume <30 ml/hr, or mental confusion); 3. need to infuse a booster drug (except dopamine <5 μg/kg/min) to maintain adequate tissue perfusion and systolic blood pressure > 90 mmHg ;

* The time from onset to the time of thrombolysis is ≤ 14 days;
* Male patients must agree to take effective contraceptive measures during treatment and at least 28 days after the end of the trial, and do not donate sperm during this period; women of childbearing age must be negative within the first 72 hours of randomization, and agree to adopt effective contraceptive measures during treatment and at least 28 days afterwards the last treatment.
* Voluntary signing of written informed consent form.

Exclusion Criteria:

* a history of hemorrhagic stroke or unexplained stroke;
* Ischemic stroke or transient ischemic attack within 3 months;
* Central nervous system damage or tumor;
* Surgery and trauma of the brain or spine within 2 months;
* Active internal bleeding within 1 month (such as gastrointestinal bleeding, hemoptysis, blood in the stool, etc.);
* High risk of bleeding: evidence or history of bleeding disorders, bleeding tendency, bleeding constitution or coagulopathy;
* oral anticoagulant (can be randomized after a certain period of time, such as oral rivaroxaban can be randomized after 1 day of elution, oral warfarin can be performed at International Normalized Ratio <2.0 random);
* 1 week after pregnancy or delivery;
* vascular puncture of the site that cannot be oppressed;
* Cardiopulmonary resuscitation within 10 days;
* Hypertension that is difficult to control (systolic blood pressure > 180 mmHg and / or diastolic blood pressure ≥ 110 mmHg);
* Liver function is grade C of Child-Pugh ;
* Infective endocarditis;
* History of aneurysms or arteriovenous malformations, or suspected aortic dissection;
* Cardiac thrombosis;
* Diabetes with hemorrhagic retinopathy or other hemorrhagic eye diseases;
* Laboratory inspection:Platelets (PLT) <90×109/L;Alanine aminotransferase (ALT) > 2.5 × ULN, aspartate aminotransferase (AST) > 2.5 ×Upper Limit of Normal (ULN);Endogenous creatinine clearance (Ccr) ≤ 50ml/min (calculated according to the Cockcroft-Gault formula);Alkaline phosphatase (ALP) > 2.0 × ULN;
* Severe cardiac insufficiency occurred in the past 6 months, New York Heart Association Heart Function Rating (NYHA classification) ≥ III;
* Participate in other clinical trials within 1 month prior to enrollment;
* Known or suspected hypersensitivity to plasminogen activator, or allergic to contrast agents, or drugs administered during the trial;
* People with mental disorders;
* Accompanied by other serious diseases that may prevent them from entering or affecting their survival, such as cancer or AIDS;
* Any disease or condition that is not suitable for intravenous thrombolysis;
* Other diseases or conditions that the investigator believes are not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
the opening rate of thrombus | 48 hours (Day 3)after injection
  The pulmonary artery occlusion index is calculated according to Qanadli scores. There are 10 segmental arteries in each pulmonary artery (3 in the upper lobes, 2 in the middle or lingual arteries, and 5 in the inferior lobes), 1 segment of arterial partial obstruction is 1 point, complete obstruction is 2 points, and the total score is divided by 40 (the total score of complete obstruction of bilateral pulmonary arteries) is the pulmonary artery obstruction index.
  Thrombus opening rate is calculated by the Qanadli CT embolization index, the formula is as follows: improvement (%) = (significant improvement cases + mild improvement cases) / overall number of cases, significant improvement = Qanadli CT embolization index decreased from baseline ≥ 75%; mild improvement = Qanadli CT embolization index decreased by ≥25% and <75% from baseline; unchanged = Qanadli CT embolization index decreased <25% from baseline; deterioration = Qanadli CT embolization index increased from baseline.

SECONDARY OUTCOMES:
Mortality and recurrence rate | within 7 days after injection
  Observe the mortality and recurrence cases within in 7 days after the injection
The incidence rates of endpoint events | within 30 days after injection
  endpoint events includes mortality, recurrent rate of symptomatic venous thromboembolism,hemodynamic deterioration or any other complications.
the ratio of right ventricular end-diastolic diameter/left ventricular end-diastolic diameter | Day 2 (24h), Day 3 (48h), Day 7, Day 30 after injection
  Compare the ratio of diameter before and after the thrombolytic therapy between two groups(low dose of rPA and high dose of rPA)
The ratio of N terminal pro B type natriuretic peptide/B-type natriuretic peptide | Day 2 (24h), Day 3 (48h), Day 7, Day 30 after injection
  Compare the ratio of diameter before and after the thrombolytic therapy between two groups(low dose of rPA and high dose of rPA)
Thrombotic load | Day 3（48h）、Day 30 after injection
  Compare the ratio before and after the injection
the opening rate of thrombus | Day 30 after injection
  calculated by Qanadli CT embolization index
the occurrence rate of adverse event | through study completion, an average of 1.5 year
  Incidence of Treatment-Emergent Adverse Events
blood pressure | through study completion, an average of 1.5 year
  both systolic and diastolic will be assessed
life signs | through study completion, an average of 1.5 year
  body temperature
pulse | through study completion, an average of 1.5 year
  the beating rate of blood through the body, which can be assessed through touching
Hemoglobin | through study completion, an average of 1.5 year
  the concentration of hemoglobin will be measured and reported in the results data table
red blood cell | through study completion, an average of 1.5 year
  number of red blood cells per unit will be measured and reported in the results data table
white blood cell | through study completion, an average of 1.5 year
  number of white blood cells per unit will be measured and reported in the results data table
platelet | through study completion, an average of 1.5 year
  number of platelet per unit will be measured and reported in the results data table

CONTACTS AND LOCATIONS:
Overall Officials: zhenguo Zhai, Doctor, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No